CLINICAL TRIAL: NCT06708858
Title: Phase Ⅱ Clinical Study of Surufatinib Combined With Gemcitabine and Cisplatin Plus Durvalumab/Pembrolizumab Regimen in the Treatment of Advanced Biliary Tract Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dai, Guanghai (Other)
Responsible Party: Sponsor-Investigator, Dai, Guanghai, chief physician, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A2024-BTC-01
Record Dates: First submitted 2024-11-11; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Advanced Biliary Tract Cancer
MeSH Terms: interventions — surufatinib; Gemcitabine; Cisplatin; durvalumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GC+IO+Surufatinib (Experimental): Surufatinib Combined With Gemcitabine and Cisplatin Plus Durvalumab/Pembrolizumab
  Interventions: Drug: Surufatinib; Drug: Gemcitabine; Drug: Cisplatin; Drug: Durvalumab; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Surufatinib — 200mg，qd，po
Drug: Gemcitabine — 1000mg/ m2, IV，d1，8，q3w
Drug: Cisplatin — 25mg/m2，IV，d1，8，q3w
Drug: Durvalumab — 1500mg，IV，d1，q3w
Drug: Pembrolizumab — 200mg，IV，d1，q3w

SUMMARY:
This phase II trial studies how well gemcitabine, cisplatin and durvalumab/Pembrolizumab and surufatinib work in treating participants with advanced Biliary Tract Cancer. The international multicenter phase III clinical study TOPAZ-1 has confirmed that durvalumab combined with gemcitabine and cisplatin can bring survival benefits to advanced BTC. Whether if adding surufatinib to a standard of care can bring addition benefit needs to be explored.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with biliary tract cancer who are clearly diagnosed by pathology, are unable to undergo radical surgery or have local/distant metastasis (allowing surgical treatment after successful transformation).
2. Have at least 1 lesion that can be measured according to RECIST v1.1 (more than 1cm on CT or MRI).
3. Have not received systematic anti-tumor therapy before.
4. Expected survival greater than 3 months;
5. Age 18-75 years old, male and female;
6. Body weight > 40kg;
7. ECOG 0-1
8. Total peripheral blood white blood cells > 2×109/L;
9. Bone marrow reserve and liver and kidney function (as demonstrated by the following laboratory tests prior to initial treatment) :

   Neutrophil absolute value ≥ 1,000/mm3; Hemoglobin > 8g/dL; Platelet count > 80,000/mm3; Glutamic pyruvic transaminase/glutamic oxalacetic transaminase < 3×ULN; Serum creatinine < 3×ULN. Total bilirubin level < 3×ULN.
10. No obvious genetic disease;
11. Liver function child-pugh A ;
12. Women of childbearing age (15 to 49 years) must undergo a pregnancy test with a negative result within 7 days before starting treatment and have effective contraception within 120 days after the last cycle of treatment.
13. The previous treatment for the tumor has ended for at least 4 weeks, and the adverse reactions of the previous treatment have basically recovered (according to the CTCAE5.0 standard ≤ Grade 1, except hair loss).
14. Voluntarily enrolled in the group and signed informed consent, followed the experimental treatment plan and visit plan, and could cooperate to observe adverse events and efficacy.

Exclusion Criteria:

1. Join another clinical study at the same time, unless it is during the follow-up period of an observational (non-interventional) or supportive care clinical study or interventional study.
2. Obstructive jaundice (bilirubin > 1.5 ULN) with inadequate biliary drainage.
3. Absolute neutrophil count (ANC) <1×109/L or platelet <80×109/L or hemoglobin < 8g/dL (based on the normal value of the clinical trial center)
4. Serum total bilirubin was 5 times higher than the upper limit of the normal reference range;
5. ALT, AST or ALP above 5 times the upper limit of the normal reference range;
6. Known active central nervous system metastatic and/or cancerous meningitis; Patients with previously treated BMS may participate provided they are stable (there is no evidence of imaging progression at least 4 weeks before the first dose of trial treatment, and any neurological symptoms have returned to baseline levels), there is no evidence of new or expanded BMS, and there is no evidence of new or expanded BMS. And no use of hormones greater than 10mg prednisone per day or equivalent for at least 14 days prior to trial treatment.
7. Toxicity of previous anticancer treatment has not returned to grade 0 or 1 level (except hair loss);
8. Uncontrolled mass pleural effusion or massive ascites
9. Organ failure; Heart: Grade III and grade IV; Liver: reached Child-Pugh liver function grade B and C; Kidney: renal failure and uremia stage; Lungs: Symptoms of severe respiratory failure; Brain: A person with a disorder of consciousness.
10. History of heart disease:

1) Patients with pre-existing arrhythmias with prolonged PR, QTc and/or QRS; 2) Acute myocardial infarction or congestive heart failure within 6 months; 3) Patients with long QT syndrome; 4) Patients who have been treated with antiarrhythmic drugs (e.g. quinidine IA, amiodarone III, sotalol); 11. Patients who have undergone major surgery within 4 weeks prior to the start of study treatment, or who expect to undergo major surgery (other than surgery for diagnostic purposes) during the study period; 12.HIV antibody positive, or have other acquired, congenital immunodeficiency diseases, or have a history of organ transplantation; 13. Uncontrolled co-morbidity, including but not limited to persistent or active infections, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina, arrhythmia, interstitial lung disease, severe chronic gastrointestinal disease with diarrhea, or mental illness/social conditions, will limit compliance with study requirements. Substantially increases the risk of developing AEs or impairs a patient's ability to give written informed consent.

14. Patients with a history of Parkinson's disease or epilepsy, or who had a history of transient ischemic attacks, stroke, or traumatic brain injury with disturbance of consciousness in the 12 months prior to the study; 15. CTCAE2 grade infection that does not respond to treatment or CTCAE grade > 2 active clinically serious infection.

16. Patients with active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection who require treatment.

17. Known or suspected prior allergy or hypersensitivity to any investigational drug or to any investigational drug excipient (duvaliumab, Sofantinib, Pabolizumab).

18. Chronic diseases requiring immunological agents or hormone therapy; 19. Women who are pregnant (positive pregnancy test before medication) or breastfeeding; 20. Participated in a non-anti-PD1 /L1 antibody based clinical trial within the past 30 days.

21. Patients with rare heritability should not participate in this clinical study.

Exit criteria

If any of the following events occur, the patient must withdraw from the study:

1. Patient voluntary withdrawal
2. Ineligibility discovered after enrollment
3. Poor compliance, failure to adhere to the protocol
4. Occurrence of adverse events (AE) or serious adverse events (SAE) where the investigator determines or the patient and family prefer not to continue treatment
5. Pregnancy
6. Inability to complete treatment according to the protocol after adjustment for grade 3/4 adverse events
7. Unforeseen, intolerable adverse reactions
8. Medical or ethical reasons impacting the continuation of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
ORR | Tumor assessments (per RECIST 1.1) every 6 weeks for the first 24 weeks and then every 8 weeks, through study completion, an average of 1 year
  Disease assessments based on investigator assessments were determined by using RECIST version 1.1 guidelines. The ORR was defined as the percentage of patients with confirmed complete response (CR) or confirmed partial response (PR). The CR was defined as disappearance of all target and non-target lesions and no new lesions. The PR was defined as >= 30% decrease in the sum of diameters of target lesions (compared to baseline) and no new non-target lesion. A confirmed CR or PR was defined as 2 CRs or 2 PRs with no evidence of progression in-between. Patients who discontinued randomized treatment without progression, received a subsequent anti-cancer therapy and then responded were not included as responders for ORR.

SECONDARY OUTCOMES:
PFS | Tumor assessments every 6 weeks for the first 24 weeks and then every 8 weeks thereafter until date of RECIST 1.1 defined radiological progressive disease or death,through study completion, an average of 1 year.
  PFS based on investigator assessments according to RECIST version 1.1 was defined as time from date of treatment until date of objective disease progression or death (by any cause in the absence of progression), regardless of whether the patient withdrew from therapy or received another anticancer therapy prior to progression. Progression (i.e., PD) was defined as at least a 20% increase in the sum of diameters of target lesions (TLs) and an absolute increase of ≥5mm, taking as reference the smallest sum of diameters since treatment started including the baseline sum of diameters, or a measurable increase in a non-target lesion, or the appearance of new lesions. Median PFS was calculated using the Kaplan-Meier technique.
OS | through study completion, an average of 24 weeks
  Overall Survival (OS) was defined as the time from the date of treatment until death due to any cause. Any patient not known to have died at the time of analysis was censored based on the last recorded date on which the patient was known to be alive. Median OS was calculated using the Kaplan-Meier technique.
conversion rate | through study completion, an average of 2 year
  Number of patients amendable to curative surgical interventions defined as number of patients receiving curative surgical resection or transplantation after successful down-sizing of tumor(s) by intervention.
safety | from the date of treatment to 90 days after last treatment
  Incidence, nature, and severity of adverse events graded according to the United States National Cancer Institute The Common Terminology Criteria for Adverse Events (NCI CTCAE 5.0)

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China